CLINICAL TRIAL: NCT05001542
Title: Could Digital Interventions Help Understand And "Flatten The Curve" Of Distress Due To Moral Injury Among Health Care Workers During The COVID Pandemic?
Brief Title: Digital Interventions for Detection and Reduction of Moral Distress
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto Metropolitan University (Other); University of Toronto (Other); University of Ontario Institute of Technology (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Venkat.Bhat, Principal Investigator, Unity Health Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-066; CPCA-0592 (Other Grant/Funding Number: DND Canada: IDEaS Competitive Projects)
Record Dates: First submitted 2021-07-28; First posted 2021-08-12 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Moral Injury; Distress, Emotional
Keywords: Depression; Anxiety; Stress; Moral Injury; Moral Distress; Loneliness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Users will go through a VR experiment before and after a brief interventional informative video describing moral distress. The VR experiment is a simulation that will lead the participant through a stressful experience about moral distress during the COVID-19 pandemic. Before, during, and after the experiment, active and physiological data will be collected from the participant to monitor their level of acute distress and health, respectively. Following the experiment, active and passive data will be collected on each user through the investigators' mobile platform (DiiG) for longitudinal monitoring of moral distress and injury.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): VR simulation exercise with a digital follow-up component to help assess the physiological and psychological indicators of moral distress
  Interventions: Other: Educational moral injury video

INTERVENTIONS:
Other: Educational moral injury video — Educational video that addresses the identification of moral injury and distress in frontline healthcare workers during COVID-19; offers available interventions at the levels of individual, team and organization

SUMMARY:
Stress, anxiety, distress and depression are exceptionally high among healthcare workers at the frontline of the COVID-19 pandemic. Factors underlying distress and resilience are unknown and there are no evidence based interventions to impact the mental wellbeing of frontline healthcare workers. This study will evaluate a novel virtual reality platform to gather the "distress experience" of frontline healthcare workers at Unity Health Toronto in real time during the ongoing COVID pandemic by developing and showing feasibility of digital technology (Virtual Reality (VR) and mobile app) as a digital platform to understand the causes and ultimately reduce the moral distress of healthcare providers during the COVID-19 pandemic. The project will develop innovations which can be used for future pandemics and other contexts prone to producing moral distress and injury.

ELIGIBILITY:
Inclusion Criteria:

* Staff or healthcare providers working at Unity Health Toronto
* 18 years of age or older
* Must own a mobile phone running Android Version 6.0 and higher, or an iPhone 6 running OS 14 and higher)

Exclusion Criterion:

- Non-Unity Health Toronto staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Feasibility evaluation of the virtual reality environment | 60 minutes (during the intervention)
  The primary outcome measure will be a comparison of MIOS (Moral Injury Outcome Scale) and PSS (Perceived Stress Scale) scores before and after watching an educational video on moral injury; feasibility of this platform will be assessed based on a feasibility questionnaire and changes in score.

SECONDARY OUTCOMES:
Feasibility evaluation of a mobile platform to understand the continuum of stress and moral distress. | Up to 8 weeks
  Feasibility of the mobile platform will be measured based on dropout rate

CONTACTS AND LOCATIONS:
Overall Officials: Venkat Bhat, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Espinola CW, Nguyen B, Torres A, Sim W, Rueda A, Beavers L, Campbell DM, Jung H, Lou W, Kapralos B, Peter E, Dubrowski A, Krishnan S, Bhat V. Digital Interventions for Stress Among Frontline Health Care Workers: Results From a Pilot Feasibility Cohort Trial. JMIR Serious Games. 2024 Jan 9;12:e42813. doi: 10.2196/42813. PMID 38194247
- [Derived] Nguyen B, Torres A, Sim W, Kenny D, Campbell DM, Beavers L, Lou W, Kapralos B, Peter E, Dubrowski A, Krishnan S, Bhat V. Digital Interventions to Reduce Distress Among Health Care Providers at the Frontline: Protocol for a Feasibility Trial. JMIR Res Protoc. 2022 Feb 16;11(2):e32240. doi: 10.2196/32240. PMID 34871178